CLINICAL TRIAL: NCT01923844
Title: Effects of Bolus Surfactant Therapy on Serial Peripheral Perfusion Index and Tissue Carbon Monoxide Measurements in Preterm Infants With Severe Respiratory Distress Syndrome
Brief Title: Effects of Bolus Surfactant Therapy on Peripheral Perfusion Index and Tissue Carbon Monoxide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Mehmet Yalaz, Attending Neonatologist, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: surf_pi_co_1
Record Dates: First submitted 2013-08-13; First posted 2013-08-16 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: Respiratory Distress Syndrome
Keywords: Newborn; perfusion index; pulsatility index; respiratory distress syndrome; surfactant; transcutaneous carbon monoxide
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — beractant

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- poractantalfa (Experimental): preterm infants who received poractantalfa for respiratory distress syndrome
  Interventions: Drug: exogenous surfactant
- beractant (Experimental): preterm infants who received beractant for respiratory distress syndrome
  Interventions: Drug: exogenous surfactant
- Control (No Intervention): Preterm infants without respiratory distress syndrome

INTERVENTIONS:
Drug: exogenous surfactant — Preparations of poractantalfa (Curosurf, 200 mg/kg) (n = 15) or beractant (Survanta, 100 mg/kg) (n = 15) were administered in a consecutive randomized manner within the first 6 h of life. During the procedure, the tube was disconnected from the ventilator. The patient's head was held in a neutral position and surfactant preparations were given in two bolus fractions. Manual ventilation was given for 2 min after each dose. After the second dose, the endotracheal tube was reconnected and the physician (D.T.) observed the infant for 30-60 s until the oxygen saturation reached > 90% on pulse oximetry. Thereafter, the peak inspiratory pressure of the 6 ventilator was reduced by 1-2 mmH2O.
  Other Names: poractantalf; beractant
  Arms: beractant; poractantalfa

SUMMARY:
Exogenous bolus surfactant administration may affect hemodynamic parameters and peripheral perfusion. Surfactant therapy is commonly used for respiratory distress syndrome in premature infants, which is also associated with inflammation. There are different types and doses of surfactant preparations available. With the help of new generation monitors, changes in peripheral perfusion and transcutaneous CO, a marker of inflammation, may be demonstrated.

DETAILED DESCRIPTION:
Preterm infants with severe Respiratory Distress Syndrome (study group) were compared to preterm infants without Respiratory Distress Syndrome(control group). Infants in the study group were randomized to receive either poractantalfa or beractant.

Perfusion index (PI) and transcutaneous CO (TCO) values were measured before (Tp) and 0 (T0), 5 (T5), 30 (T30), 60 (T60), 360 (T360) minutes after surfactant administration in the first six hours of life.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 26 and 36 weeks
* intubated for respiratory distress syndrome

Exclusion Criteria:

* cardiac defects,
* hemodynamically significant patent ductusarteriosus,
* congenital pneumonia,
* early sepsis
* unstable infants in need of inotropic support.

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in perfusion index (PI)at 6 hours | before (Tp) and 0 (T0), 5 (T5), 30 (T30), 60 (T60), 360 (T360) minutes after surfactant administration in the first six hours of life
  PI values were measured before (Tp) and 0 (T0), 5 (T5), 30 (T30), 60 (T60), 360 (T360) minutes after surfactant administration in the first six hours of life.
Change from baseline in transcutaneous carbon monoxide (TCO)at 6 hours | before (Tp) and 0 (T0), 5 (T5), 30 (T30), 60 (T60), 360 (T360) minutes after surfactant administration in the first six hours of life
  TCO values were measured before (Tp) and 0 (T0), 5 (T5), 30 (T30), 60 (T60), 360 (T360) minutes after surfactant administration in the first six hours of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Yalaz, M.D., Principal Investigator — Ege University Faculty of Medicine, Department of Pediatrics, Division of Neonatology
Locations (1):
- Ege University Children's Hospital Neonatal Intesive Care Unit, Izmir, İzmir, Turkey (Türkiye)